CLINICAL TRIAL: NCT06179485
Title: Effect of Ketamine and Etomidate During Rapid Sequence Intubation on Long- Term Outcomes (Long-Term Outcomes of the RSI Trial)
Brief Title: Effect of Ketamine and Etomidate During RSI on Long Term Outcomes
Acronym: RSI-LTO
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Assistant Professor of Medicine, Department of Medicine, Allergy, Pulmonary and Critical Care Medicine, Vanderbilt University Medical Center
Other Study IDs: 210500-2; BPS-2022C3-30021 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2023-12-08; First posted 2023-12-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Post-Traumatic Stress Disorder; Acute Respiratory Failure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Etomidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comparator: Ketamine Group: Intravenous ketamine as the sedative for induction of anesthesia during emergency tracheal intubation.
  Interventions: Drug: Ketamine
- Comparator: Etomidate Group: Intravenous etomidate as the sedative for induction of anesthesia during emergency tracheal intubation.
  Interventions: Drug: Etomidate

INTERVENTIONS:
Drug: Ketamine — The RSI-LTO study collects long-term outcomes from the RSI trial (NCT05277896). In the RSI trial, patients in the ketamine group will be assigned to receive intravenous ketamine for induction of anesthesia during tracheal intubation. A dose of 2 mg/kg will be recommended, and the group assignment sheet will contain a nomogram providing the recommended dose for a range of patient weights (in pounds and kg). Treating clinicians will be able elect to give a lesser or greater dose of ketamine than recommended if felt to be required for optimal patient care.
  Groups: Comparator: Ketamine Group
Drug: Etomidate — The RSI-LTO study collects long-term outcomes from the RSI trial (NCT05277896). In the RSI trial, patients in the etomidate group will be assigned to receive intravenous etomidate for induction of anesthesia during tracheal intubation. A dose of 0.3 mg/kg will be recommended, and the group assignment sheet will contain a nomogram providing the recommended dose for a range of patient weights (in pounds and kg). Treating clinicians will be able elect to give a lesser or greater dose of etomidate than recommended if felt to be required for optimal patient care.
  Groups: Comparator: Etomidate Group

SUMMARY:
The RSI-LTO study collects long-term outcomes from the RSI trial (NCT05277896). One-third of adults who are intubated in the ED or ICU experience symptoms of posttraumatic stress disorder (PTSD). PTSD is a psychiatric disorder triggered by a "shocking, scary, or dangerous event." Critical illness, tracheal intubation, and mechanical ventilation can be traumatic and distressing events. Patients may recall the intubation procedure, the feeling of the breathing tube in their throat, or being unable to move ("paralyzed"). While on the breathing machine, patients may experience delirium, frightening hallucinations, and delusions. Patients with PTSD after critical illness can be hypervigilant, anxious, and troubled by intrusive thoughts, nightmares, and flashbacks that last months to years after critical illness and that PTSD negatively impacts patients' marriages, work, and quality of life and increases patients' risk of depression, anxiety, substance use disorder, and suicide. Ketamine may prevent PTSD symptoms by blocking the pathways in the brain's glutaminergic system that are responsible for the formation of traumatic memories In outpatients with chronic PTSD, a single dose of ketamine has been shown to reduce PTSD symptoms for up to 2 weeks. Even a modest reduction in PTSD would translate into tens of thousands of fewer cases of PTSD each year, more cases of PTSD each year than any other medical intervention evaluated to date.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in RSI trial (NCT05277896)

Exclusion Criteria:

* Aphasic or non-verbal prior to tracheal intubation
* Cannot follow commands prior to tracheal intubation
* Non-English speaking
* Deaf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults undergoing emergency tracheal intubation who were enrolled in the RSI trial (NCT05277896) and meet eligibility criteria for long-term outcomes assessment.
Sampling Method: Non-Probability Sample
Enrollment: 1756 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptoms at 12 months | 12 months
  The investigators will measure PTSD symptoms at 3 and 12 months using the Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5). The PCL-5 is a widely used 5-10 minute patient survey validated to characterize severity of symptoms of PTSD. Patients rate 20 items corresponding to the DSM-5 criteria for PTSD on a 5-point Likert scale ranging from 0 (not bothersome) to 4 (extremely bothersome). Total scores range from 0 to 80, with higher scores indicating more severe symptoms of PTSD. Because a value for the PCL-5 score will not exist for patients who die prior to assessment, the main analysis will use a composite endpoint approach where patients whose PCL-5 could not be assessed because they died will be assigned a value of 81 (higher than the worst value on the PTSD symptom scale).

OTHER OUTCOMES:
Vital status | 12 months
  Date and location of death will be assessed from enrollment until 12 months after enrollment by trial personnel using review of electronic health records, phone calls with families, and national death indices.
Awareness of paralysis | 3 months
  This will be determined by the modified Brice questionnaire and ICU Memory Tool (15-20 minutes). These semi-structured interviews ask subjects about their recollection of the ICU experience, including of being paralyzed. Possible awareness with paralysis event (Present/Absent) will be defined as: (1)reporting memories of the period between losing consciousness and waking up and (2) a sensation/feeling of wakeful paralysis.
ICU Memories | 3 months
  This will be determined by the ICU Memory Tool (15-20 minutes). These semi-structured interviews ask subjects about their recollection of the ICU experience, including emotions, memories, and the worst thing experienced during mechanical ventilation. Patients will be classified as having (1) factual memories, (2) delusional memories, (3) memories of feelings. These choices are not mutually exclusive as they may have more than one or none of these memories.
Threat perception | 3 months
  This 7-item questionnaire assesses the patient's perception of feeling threatened during the intubation experience. Scores range from 0 (none at all) to 21 (extremely threatened).
Anxiety | 12 months
  Anxiety symptoms will be characterized using the General Anxiety Disorder-7 (GAD-7) which is a 7-item questionnaire that ranges from 0 (no anxiety) to 21 (severe anxiety).
Depression | 12 months
  Depression symptoms will be characterized using the Patient Health Questionnaire-9 (PHQ-9) which is a 9-item questionnaire that ranges from 0 (no depression) to 27 (severe depression).
Quality of life (EQ-5D-5L) | 12 months
  Quality of life will be characterized using the EuroQol 5-Dimension, 5 level version (EQ-5D-5L) is a 5-question instrument that captures impairments in mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. EQ-5D-5L scores will be summarized using the index value validated for the US population. Index scores range range from -0.573 (quality of life worse than death) to 1.000 (perfect quality of life).
Global Cognition | 12 months
  Global cognition will be characterized using the Montreal Cognitive Assessment - Blind (MoCA-Blind). The MoCA-Blind assesses memory, attention, language, abstraction, delayed recall, and orientation. Scores range from 0 (severe cognitive impairment) to 22 (no cognitive impairment).
Executive Function | 12 months
  Oral Trailmaking Test - Patient counts from 1 to 25 and then alternates between numbers and letters (i.e., 1-A-2-B-3-C, etc.,)
Loss of Employment | 12 months
  Patients are asked what their employment status is prior to the acute illness and at 12-months. Patients will be considered to be have loss of employment if they go from: (1) full to partial employment, (2) full to no employment, or (3) partial to no employment.
Physical disability | 12 months
  Duke Activity Status Index (DASI) - An 11-item survey that assesses the patient's current ability to perform various physical activities. Scores range from 0 (poor physical function) to 58.2 (excellent physical function).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of Colorado Denver, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Following publication, individual patient data will be made available for sharing to researchers with 1) a signed data access agreement, 2) research testing a hypothesis, 3) a protocol that has been approved by an institutional review board, and 4) a proposal that has received approval from the principal investigator.
Supporting Information: Study Protocol, SAP, ICF